CLINICAL TRIAL: NCT07067853
Title: Effectivity and Safety of GB20 Acupoint Pharmacopuncture With Lidocaine 2% on Migraine Patients : Study on Head Pain Characteristic and MIDAS-Ina Score
Brief Title: Effectivity and Safety of GB20 Acupoint Pharmacopuncture With Lidocaine 2% on Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Jeffry Alamsjah, Principal Inverstigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 25-07-0995
Record Dates: First submitted 2025-07-14; First posted 2025-07-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: Migraine; Acupuncture
MeSH Terms: conditions — Migraine Disorders | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: The intervention group will receive pharmacopuncture, while the control group will receive propranolol tablets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Injection of 0.5mL Lidocaine 2% solution into GB20 acupuncture point, both sides every week for 4 week
  Interventions: Device: Lidocaine 2 % Pharmacopuncture
- Control Group (Active Comparator): Propranolol 20mg, twice daily for 28 day / 4 week
  Interventions: Drug: propranolol 20mg

INTERVENTIONS:
Device: Lidocaine 2 % Pharmacopuncture — Injection of 0.5mL Lidocaine 2% solution into GB20 acupuncture point, both sides every week for 4 week
  Arms: Intervention Group
Drug: propranolol 20mg — Propranolol 20mg, twice daily for 28 day / 4 week
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if 2% Lidocaine pharmacopuncture at the GB20 acupoint can effectively and safely treat migraine in adult patients. The main questions it aims to answer are:

* Does 2% Lidocaine pharmacopuncture at GB20 reduce the frequency of migraine attacks more than 40mg propranolol?
* Does 2% Lidocaine pharmacopuncture at GB20 reduce the duration of migraine attacks more than 40mg propranolol?
* Does 2% Lidocaine pharmacopuncture at GB20 reduce the intensity of migraine pain more than 40mg propranolol?
* Does 2% Lidocaine pharmacopuncture at GB20 improve MIDAS-Ina scores more than 40mg propranolol?
* Is 2% Lidocaine pharmacopuncture at GB20 more effective in improving bothersome migraine symptoms compared to 40mg propranolol?
* What is the incidence of side effects of 2% Lidocaine pharmacopuncture at GB20 in migraine patients?

Researchers will compare a pharmacopuncture group to a conventional medication group (propranolol) to see if pharmacopuncture works as an effective and safe alternative treatment for migraine patients.

Participants will:

* In the pharmacopuncture group, receive weekly injections of 0.5cc of 2% Lidocaine at the GB20 acupoint (bilaterally) for four weeks. These injections will be guided by ultrasonography.
* In the medication group, receive 20mg propranolol tablets twice daily for 28 days.
* Be provided with 500mg Paracetamol tablets as abortive therapy for acute migraine attacks.
* Use the 'Guardian Headache Diary' application to record migraine attack data (frequency, duration, intensity) for two months.
* Complete the MIDAS-Ina questionnaire at the beginning of the study, at the end of week 4, and at the end of week 8.

Side effects will be monitored and recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with migraine
* Minimum of 3 days of migraine attacks in 1 month
* Willing to participate until the study concludes

Exclusion Criteria:

* Headache with other known cause (e.g. head trauma, cancer, hemorrhagic stroke)
* Inaccessible GB20 acupuncture point (scar tissue, infection, open wound, etc)
* History of heart disease and/or asthma
* History of Hypersensitivity with propranolol and/or lidocaine
* History of acupuncture treatment 3 month prior to study
* Routine consumption of anticoagulation medications, steroids or pain killers
* Pregnant and breastfeeding women

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Frequency of migraine attacks | Before therapy, week 4, week 8
  Frequency of migraine attacks in 1 month
Duration of migraine attacks | Before therapy, week 4, week 8
  Duration of migraine attacks, counted in hour
Intensity of migraine attacks | Before therapy, week 4, week 8
  intensity of migraine attacks, measured with numeric rating scale from 1 to 10
Migraine Disability Assessment Test - Indonesian Language (MIDAS-Ina) Score | Before therapy, week 4, week 8
  Disability caused by migraine will be assessed with Migraine Disability Assessment Test - Indonesian Language (MIDAS-Ina), a 5-question questionnaire with a minimum score of 0 and maximum score of 450. Higher score means worse outcome.
Bothersome Symptom Improvement | week 4, week 8
  Improvement of bothersome symptoms, measured as improved or not improved
Adverse Event Related to Intervention | immediately post-intervention until 8 weeks
  adverse event happening after intervention is given, including pain, infection, skin rash/irritation will be recorded and monitored

CONTACTS AND LOCATIONS:
Overall Officials: Komite Etik Penelitian Kesehatan FKUI-RSCM, Principal Investigator — Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided